CLINICAL TRIAL: NCT02069236
Title: Correlation of G6PD Activity Across Different Sample Sources, and Different G6PD Testing Platforms
Brief Title: Comparing G6PD Tests Using Capillary Blood Versus Venous Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Mahidol University (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SMRU 1302
Record Dates: First submitted 2014-02-14; First posted 2014-02-24 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2014-02

CONDITIONS: Glucose-6 Phosphate Dehydrogenase Deficiency
Keywords: Glucose-6 phosphate dehydrogenase deficiency; capillary; venous; genotype phenotype correlation
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency | interventions — Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G6PD Testing (No Intervention): All subjects receive G6PD test
  Interventions: Other: G6PD Test

INTERVENTIONS:
Other: G6PD Test — All subjects are tested by multiple G6PD tests
  Other Names: Trinity spectrophotometric assay; Flow cytometry; CareStart; Florescent Spot Test

SUMMARY:
In this study we propose to determine the correlation in glucose-6phosphate dehydrogenase enzyme activity in capillary blood obtained from a finger stick versus a venous blood specimen. As secondary endpoints we will seek to correlate phenotype as determined by quantitative and qualitative G6PD test, genotype as determined by PCR and DNA sequencing with flow cytometry. The secondary endpoints are critical for the design of G6PD diagnostic test evaluation studies.

DETAILED DESCRIPTION:
In this study we propose to determine the correlation in glucose-6 phosphate dehydrogenase enzyme activity in capillary blood obtained from a finger stick versus a venous blood specimen. We will also compare results of different G6PD tests with known G6PD genetic profiles. The results of the study will inform design of future G6PD diagnostic development & evaluations. This research will be conducted in MaeSot Thailand, where G6PD deficiency has a high prevalence. Study participants will be recruited into three groups of 50 volunteers per group: 50 G6PD-deficient individuals, 50 G6PD-normal individuals, and 50 G6PD-intermediate individuals. Following a written informed consent, participants will donate about 3 ml of venous blood and about 4 drops of capillary blood (fingerstick). There will be no direct benefit to research participants.

ELIGIBILITY:
Inclusion Criteria:

* Previous G6PD test at SMRU clinic
* Patient willing to participate and sign informed consent form
* Patient willing to allow donated sample to be used in future research
* Subjects 18 years of age or older

Exclusion Criteria:

* patients with severe malaria or other severe illness
* Patients who received a blood transfusion in the last 3 months
* Patients who received primaquine in the past 1 month (this is to ensure that previous characterization of phenotype in the healthy subject has not been influenced by a recent hemolytic reaction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Correlation of capillary and venous blood results using Trinity quantitative G6PD test | Six months
  Comparison of the performance of the Trinity quantitative test using capillary blood, vs the performance of the same test using venous blood.

SECONDARY OUTCOMES:
Concordance between a flow cytometry-based G6PD test and the spectrophotometric gold standard | six months
  Percent agreement between the quantitative results of the flow cytometry assay and the quantitative results of the spectrophotometric assay.
Categorical accuracy of a flow cytometry-based G6PD test against the spectrophotometric gold standard and genotyping | six months
  Using a predefined cutoff to categorize values from each quantitative test, determine percent agreement within each category between the two tests.
Concordance between a qualitative G6PD test and the spectrophotometric gold standard | Six months
  Compare sensitivity & specificity of qualitative results of the G6PD test and the categorical results of the quantitative spectrophotometric assay.
Categorical accuracy of qualitative G6PD test against spectrophotometric gold standard | six months
  Percent agreement between the qualitative G6PD test and the categorical results of the spectrophotometric gold standard
Association between flow cytometry-based test and sample genotype | Six months
  Determine accuracy of phenotypic results of flow cytometry assay against genetic profile.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Nosten, MD/PhD, Principal Investigator — Shoklo Malaria Research Unit, Mahidol Oxford Research unit; Gonzalo Domingo, PhD, Study Chair — PATH; Germana Bancone, PhD, Study Chair — Shoklo Malaria Research Unit, Mahidol Oxford Research unit; Sarah McGray, MPH, Study Chair — PATH
Locations (1):
- Shoklo Malaria Research Unit (SMRU), Mae Sot, Thailand